CLINICAL TRIAL: NCT00333034
Title: A Multicenter, Parallel, Randomized, Double-Blind, Placebo-Controlled Trial Evaluating the Safety and Efficacy of Etanercept 50 mg Once Weekly in Subjects With Moderate to Severe Plaque Psoriasis
Brief Title: Study Evaluating the Safety and Efficacy of Etanercept 50 mg Once Weekly in Subjects With Psoriasis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Wyeth is now a wholly owned subsidiary of Pfizer (Industry)
Collaborators: Amgen (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 0881A6-318
Record Dates: First submitted 2006-05-23; First posted 2006-06-02 (Estimated); Last update posted 2007-12-06 (Estimated); Status verified 2007-12

CONDITIONS: Psoriasis
Keywords: Psoriasis
MeSH Terms: conditions — Psoriasis | interventions — Etanercept

INTERVENTIONS:
Drug: Etanercept

SUMMARY:
The primary objective is to assess the efficacy and safety of etanercept 50 mg administered once weekly in subjects with psoriasis over 12 weeks.

ELIGIBILITY:
Inclusion Criteria: -Adults greater than or equal to 18 years of age with clinically stable plaque psoriasis involving greater than or equal to 10% of the body surface and a minimum Psoriasis Area and Severity Index (PASI) score of 10 at screening. -Failure to respond to, or have a contraindication to, or intolerant to at least 1 of the following systemic or phototherapies at an adequate dose of sufficient duration: Methotrexate (MTX), Acitretin, Cyclosporine, Ultraviolet A (UVA), Ultraviolet B (UVB), Psoralen and Ultraviolet A (PUVA), Fumarate Exclusion Criteria: -Previous treatment with etanercept, antibody to TNF or other TNF inhibitors. -Active guttate, erythrodermic, or pustular psoriasis at the time of the screening or baseline.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2006-06; Study Completion 2007-05 (Actual)

PRIMARY OUTCOMES:
The primary efficacy endpoint is the PASI 75 response at week 12. PASI 75 is defined as a 75% or greater improvement in PASI score from baseline.

SECONDARY OUTCOMES:
The secondary efficacy endpoints will include but not limited to: PASI 50, PASI 75 (at visit other than week 12, PASI 90, PASI score PGA of 0 or 1 (clear or minimal, Patient global assessment of psoriasis, DLQI,
EQ5D, FACIT-F.

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Wyeth is now a wholly owned subsidiary of Pfizer; Trial Manager, Principal Investigator — For Austria, medinfo@wyeth.com; Trial Manager, Principal Investigator — For Belguim, trials-BEL@wyeth.com; Trial Manager, Principal Investigator — For France, infomedfrance@wyeth.com; Trial Manager, Principal Investigator — For Germany, medinfoDEU@wyeth.com; Trial Manager, Principal Investigator — For Hungary, WPBUMED@wyeth.com; Trial Manager, Principal Investigator — For Italy, descresg@wyeth.com; Trial Manager, Principal Investigator — For Netherlands, trials-NL@wyeth.com; Trial Manager, Principal Investigator — For Poland, WPWZMED@wyeth.com; Trial Manager, Principal Investigator — For Romania, WVPIMED@wyeth.com; Trial Manager, Principal Investigator — For Spain, infomed@wyeth.com
Locations (22):
- Innsbruck, Austria
- Belgium (2):
  - Brussels
  - Leuven
- Paris, France
- Germany (5):
  - Bonn
  - Hamburg
  - München
  - Münster
  - Regensburg
- Hungary (2):
  - Miskolc
  - Szolnok
- Italy (2):
  - Messina
  - Novara
- Netherlands (2):
  - Drachten
  - Nijmegen
- Poland (2):
  - Lodz
  - Wroclaw
- Romania (2):
  - Bucharest
  - Cluj-Napoca
- Spain (3):
  - A Coruña
  - Madrid
  - Seville

REFERENCES:
- [Derived] Griffiths CE, Christophers E, Szumski A, Jones H, Mallbris L. Impact of early vs. late disease onset on treatment response to etanercept in patients with psoriasis. Br J Dermatol. 2015 Nov;173(5):1271-3. doi: 10.1111/bjd.13865. Epub 2015 Aug 17. No abstract available. PMID 25913550